CLINICAL TRIAL: NCT04345523
Title: Multi-center, Randomized Clinical Trial of Convalescent Plasma Therapy Versus Standard of Care for the Treatment of COVID-19 in Hospitalized Patients
Brief Title: Convalescent Plasma Therapy vs. SOC for the Treatment of COVID-19 in Hospitalized Patients
Acronym: ConPlas-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cristina Avendaño Solá (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor-Investigator, Cristina Avendaño Solá, MD, PhD, Puerta de Hierro University Hospital
Organization: Puerta de Hierro University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ConPlas-19
Record Dates: First submitted 2020-04-02; First posted 2020-04-14 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: COVID-19
Keywords: COVID-19; Coronavirus; SARS-CoV-2; Convalescent Plasma; SOC; CP
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Blood Specimen Collection; Standard of Care

STUDY DESIGN:
Intervention Model Description: 1:1 ratio for CP: Control arm. Also, approximately 140-200 CP donors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Experimental): Pathogen-reduced CP from patients recovered from COVID-19, whom, for the purpose of this trial, are herein designated as donors.
  Interventions: Other: Blood and derivatives.
- Control Arm (Active Comparator): Standard of Care (SOC) for COVID-19
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Other: Blood and derivatives. — Administration of fresh plasma from donor immunized against COVID-19
  Other Names: Convalescent Plasma from patients recovered from COVID-19
  Arms: Treatment Arm
Drug: Standard of Care — Standard of care for the treatment of COVID-19 in hospitalized patients
  Other Names: SOC
  Arms: Control Arm

SUMMARY:
A total of 278 patients are planned.

All patients will be in an early-stage of COVID-19. They must be adults and hospitalized.

In this study, all participating patients will receive the standard treatment provided according to the current treatment protocols for coronavirus disease. In addition to this treatment, each patient will be randomly assigned to receive additional treatment with convalescent plasma transfusion (CP; blood plasma from patients who have been cured of coronavirus), or continue with standard treatment but without adding transfusion.

50% of the chances of additional treatment with CP, and 50% of the chances of receiving only the standard treatment for coronavirus.

The duration of the study shall be one month from the assignment of the treatment.

The patient and the doctor will know the treatment assigned.

DETAILED DESCRIPTION:
A multi-center, randomized, clinical trial with two arms to study the efficacy and safety of passive immunotherapy with CP compared to a control of standard of care (SOC).

All trial participants will receive SOC:

* Treatment arm: Pathogen-reduced CP from patients recovered from COVID-19, whom, for the purpose of this trial, are herein designated as donors.
* Control arm: SOC for COVID-19.

Randomization among the two arms will be 1:1 and will be stratified per center. Of note, in the current status of a worldwide pandemic for which we have no approved vaccines or drugs, for the purpose of this trial SOC would also accept any drugs that are being used in clinical practice (e.g. lopinavir/ritonavir; darunavir/cobicistat; hydroxy/chloroquine, tocilizumab, etc.), other than those used as part of another clinical trial.

The study is planned with a sequential design. Interim analyses: comprehensive safety data monitoring analyses will be conducted when 20%, 40%, 60% and 80% of patients, or at the discretionary DSMB criteria when needed. A DSMB charter will be set before the trial initiation where criteria for prematurely stopping the trial due to safety issues will be set. Interim analyses will be predefined upfront based on the DSMB recommendations.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to performing study procedures. Witnessed oral consent will be accepted in order to avoid paper handling. Written consent by patient or representatives will be obtained as soon as possible.
2. Male or female adult patient ≥18 years of age at time of enrolment.
3. Has laboratory-confirmed SARS-CoV-2 infection as determined by PCR in naso/oropharyngeal swabs or any other relevant specimen in the ongoing COVID-19 symptomatic period. Alternative test (i.e antigenic tests) are also acceptable as laboratory confirmation if their adequate specificity has been accepted by the sponsor.
4. Patients requiring hospitalization for COVID-19 without mechanical ventilation (invasive or non-invasive) or high flow oxygen devices and at least one of the following:

   * Radiographic evidence of pulmonary infiltrates by imaging (chest x-ray, CT scan, etc.), OR
   * Clinical assessment (evidence of rales/crackles on exam) AND SpO2 ≤ 94% on room air that requires supplemental oxygen.
5. No more than 7 days between the onset of symptoms (fever or cough) and treatment administration day.

Exclusion Criteria:

1. Requiring mechanical ventilation (invasive or non-invasive) or high flow oxygen devices.
2. More than 7 days since symptoms (fever or cough).
3. Participation in any other clinical trial of an experimental treatment for COVID-19.
4. In the opinion of the clinical team, progression to death is imminent and inevitable within the next 24 hours, irrespective of the provision of treatments.
5. Any incompatibility or allergy to the administration of human plasma.
6. Stage 4 severe chronic kidney disease or requiring dialysis (i.e. eGFR <30).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2020-04-03 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2021-04-05 (Actual)

PRIMARY OUTCOMES:
Category Changes in the "7-Ordinal Scale" | 15 days
  Proportion of patients in categories 5, 6 or 7 of the 7-point ordinal scale at day 15 7- Ordinal scale:
  1. Not hospitalized, no limitations on activities.
  2. Not hospitalized, limitation on activities.
  3. Hospitalized, not requiring supplemental oxygen.
  4. Hospitalized, requiring supplemental oxygen.
  5. Hospitalized, on non-invasive ventilation or high flow oxygen devices.
  6. Hospitalized, on invasive mechanical ventilation or ECMO.
  7. Death.

SECONDARY OUTCOMES:
Status at day 30 in the "7-point ordinal scale" | 30 days
  Status at day 30 in the "7-point ordinal scale"
Time to category 5, 6 or 7 of the " 7-Ordinal scale" | 29 days
  Time to change from baseline category to worsening into 5,6 or 7 categories of the "7-Ordinal scale"
Time to an improvement of one category from admission in the "7-Ordinal scale" | 29 days
  Time to an improvement of one category from admission in the "7-Ordinal scale"
Time to first deterioration | 60 days
  Time to first deterioration
Mean change in the ranking in the "7-Ordinal scale" from baseline to days 3,5,8,11,15,29 and 60 | 60 days
  Mean change in the ranking in the "7-Ordinal Scale" from baseline to days 3,5,8,11,15,29 and 60
Mean change in the ranking in the "11-Ordinal scale from baseline to days 3,5,8,11,15,29 and 60. | 60 days
  Mean change in the ranking in the "11- Ordinal scale" from baseline to days 3,5,8,11,15,29 and 60.
Status at day 15 and 30 in the "11-Ordinal scale" | 30 days
  Status at day 15 and 30 in the "11-Ordinal scale"
  Status at day 15 and 30 in the "11-Ordinal scale"
Mortality of any cause at 15 days | 15 days
  Rate of mortality of any cause within first 15 days.
Mortality of any cause at 28 days (day 29) | 28 days (day 29)
  Rate of mortality of any cause within first 28 days.
Mortality of any cause at 60 days | 60 days
  Rate of mortality of any cause within first 60 days.
Oxygenation free days | 29 days
  days free from oxygen supplementation
Ventilator free days | 29 days
  days free from mechanical ventilation
Duration of hospitalization (days) | 60 days
  days of hospitalization
Incidence of thrombotic arterial events | 60 days
  incidence of thrombotic arterial events
Incidence of thrombotic venous events | 60 days
  incidence of thrombotic venous events
Status at day 30 in the "11-Ordinal scale" | 30 days
  Status at day 30 in the "11-Ordinal scale"
  "11-Ordinal scale" :
  0. Uninfected ; no viral RNA detected.
  1. Asymptomatic; viral RNA detected, limitation on activities.
  2. Symptomatic; independent
  3. Symptomatic; assistance needed
  4. Hospitalized, no oxygen therapy.
  5. Hospitalized, oxygen by mask or nasal prongs
  6. Oxygen by mask or nasal prongs
  7. Intubation and mechanical ventilation, pO2/FiO2 ≥150 or SpO2/FiO2 ≥200
  8. Mechanical ventilation pO2/FIO2 <150 (SpO2/FiO2 <200) or vasopressors
  9. Mechanical ventilation pO2/FiO2 <150 and vasopressors, dialysis, or ECMO
  10. Dead
Infusion-related adverse events | 60 days
  Infusion-related adverse events Cumulative incidence of serious adverse events (SAEs) Cumulative incidence of Grade 3 and 4 adverse events (AEs).
Incidence of Treatment-Emergent Adverse Events | 60 days
  cumulative incidence of Grade 3 and 4 adverse events (AEs) Cumulative incidence of serious adverse events (SAEs) Cumulative incidence of Grade 3 and 4 adverse events (AEs).
rate of rehospitalizations | 60 days
  rehospitalizations
Antibodies levels in CP donors recovered from COVID-19 | 3 months
  Quantitative total antibodies and neutralizing antibody activity against SARSCoV-2 in the sera from donors and patients using viral pseudotypes
Viral load | Days 1,3,5,8,11,15, 29 and 60
  Change in PCR for SARS-CoV-2 in naso/oropharyngeal swabs at baseline and at discharge
Viral load | Days 1,3,5,8,11,15,29 and 60
  Change in PCR for SARS-CoV-2 in blood on Days 3,5,8,11,15,29 and 60 (while hospitalized) until two of them are negative consecutively

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Avendaño Solá, MD, PhD, Study Chair — Hospital Universitario Puerta de Hierro Majadahonda; Rafael Duarte Palomino, MD, PhD, Study Chair — Hospital Universitario Puerta de Hierro Majadahonda; Antonio Ramos, MD, PhD, Principal Investigator — Hospital Universitario Puerta de Hierro Majadahonda; José Luis Bueno, MD, Principal Investigator — Hospital Universitario Puerta de Hierro Majadahonda; Inmaculada Casas Flecha, PharmD, PhD, Principal Investigator — Centro Nacional de Microbiología, Instituto de Salud Carlos III
Locations (29):
- Spain (29):
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza, Aragon
  - Hospital Universitario Mútua Terrassa, Terrassa, Barcelona
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital General de Albacete, Albacete
  - Hospital del Mar, Barcelona
  - Hospital General Universitario de Ciudad Real, Ciudad Real
  - Hospital Universitario Donostia, Donostia / San Sebastian
  - Hospital Doctor Josep Trueta, Girona
  - Hospital Doctor Negrín, Las Palmas
  - Complejo Asistencial Universitario de León, León
  - Hospital Universitario Arnau de Vilanova, Lleida
  - Hospital San Pedro, Logroño
  - Hospital Universitario La Princesa, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Sant Joan de Deu de Manresa. Fundación Althaia, Manresa
  - Hospital Universitario de Asturias, Oviedo
  - Hospital Universitario Son Espases, Palma de Mallorca
  - Clínica Universidad de Navarra (CUN). Sedes Pamplona y Madrid, Pamplona
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Complejo Hospitalario de Toledo, Toledo
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
PD that underlie the results reported in this article, after deidenficiation (text, tables, figures, and appendices) will be shared. The data will be available after main report is published.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request.

REFERENCES:
- [Derived] Iannizzi C, Chai KL, Piechotta V, Valk SJ, Kimber C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Jindal A, Cryns N, Estcourt LJ, Kreuzberger N, Skoetz N. Convalescent plasma for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2023 May 10;5(5):CD013600. doi: 10.1002/14651858.CD013600.pub6. PMID 37162745
- [Derived] Iannizzi C, Chai KL, Piechotta V, Valk SJ, Kimber C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Jindal A, Cryns N, Estcourt LJ, Kreuzberger N, Skoetz N. Convalescent plasma for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2023 Feb 1;2(2):CD013600. doi: 10.1002/14651858.CD013600.pub5. PMID 36734509
- [Derived] Avendano-Sola C, Ramos-Martinez A, Munez-Rubio E, Ruiz-Antoran B, Malo de Molina R, Torres F, Fernandez-Cruz A, Calderon-Parra J, Payares-Herrera C, Diaz de Santiago A, Romera-Martinez I, Pintos I, Lora-Tamayo J, Mancheno-Losa M, Paciello ML, Martinez-Gonzalez AL, Vidan-Estevez J, Nunez-Orantos MJ, Saez-Serrano MI, Porras-Leal ML, Jarilla-Fernandez MC, Villares P, de Oteyza JP, Ramos-Garrido A, Blanco L, Madrigal-Sanchez ME, Rubio-Batlles M, Velasco-Iglesias A, Pano-Pardo JR, Moreno-Chulilla JA, Muniz-Diaz E, Casas-Flecha I, Perez-Olmeda M, Garcia-Perez J, Alcami J, Bueno JL, Duarte RF; ConPlas-19 Study Group. A multicenter randomized open-label clinical trial for convalescent plasma in patients hospitalized with COVID-19 pneumonia. J Clin Invest. 2021 Oct 15;131(20):e152740. doi: 10.1172/JCI152740. PMID 34473652
- [Derived] Piechotta V, Iannizzi C, Chai KL, Valk SJ, Kimber C, Dorando E, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Estcourt LJ, Skoetz N. Convalescent plasma or hyperimmune immunoglobulin for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2021 May 20;5(5):CD013600. doi: 10.1002/14651858.CD013600.pub4. PMID 34013969
- [Derived] Diago-Sempere E, Bueno JL, Sancho-Lopez A, Rubio EM, Torres F, de Molina RM, Fernandez-Cruz A, de Diego IS, Velasco-Iglesias A, Payares-Herrera C, Flecha IC, Avendano-Sola C, Palomino RD, Ramos-Martinez A, Ruiz-Antoran B. Evaluation of convalescent plasma versus standard of care for the treatment of COVID-19 in hospitalized patients: study protocol for a phase 2 randomized, open-label, controlled, multicenter trial. Trials. 2021 Jan 20;22(1):70. doi: 10.1186/s13063-020-05011-9. PMID 33472681